CLINICAL TRIAL: NCT01174147
Title: Brazilian Network of Candidemia: a Laboratory-based Surveillance Study on Candida Bloodstream Infections in 10 Medical Centers
Brief Title: A Laboratory-based Surveillance Study of Candida Bloodstream Infections (MK-0991-093)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Sponsor
Other Study IDs: 0991-093
Record Dates: First submitted 2010-07-30; First posted 2010-08-03 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Candidemia
MeSH Terms: conditions — Candidemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Hospital Candida Cases: People who developed a positive blood culture for Candida while hospitalized

SUMMARY:
This study will evaluate the incidence rate of Candida blood stream infection (candidemia) among people hospitalized in participating medical centers in Brazil, and will assess the antifungal drug susceptibility patterns of Candida clinical isolates. No hypotheses will be tested in the study. Candida blood stream isolates collected from people hospitalized for any reason during the study period will be sent to a core mycology laboratory for antifungal drug susceptibility testing. All people who develop candidemia while hospitalized will be considered participants in the study.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in a participating medical center
* Developed candidemia blood stream infection (confirmed by isolation of Candida species from blood culture)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric patients hospitalized in participating medical centers (tertiary care hospitals) in Brazil
Sampling Method: Non-Probability Sample
Enrollment: 436 (Actual)
Dates: Start 2010-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with Candidemia per 1000 hospital admissions | Approximately 1 year
  A candidemia case was defined as the first isolation of any Candida species from blood within a 30-day period during hospitalization. The incidence of candidemia was calculated as (number of participants / [number of total people hospitalized during the study period / 1000])
Number of participants with Candidemia per 1000 patient-Days in hospital | Approximately 1 year
  A candidemia case was defined as the first isolation of any Candida species from blood within a 30-day period during hospitalization. The incidence of candidemia was calculated as (number of participants / [number of total patient-days of hospitalization during the study period / 1000]).
Percentage of Specific Candida Isolates Susceptible to Amphotericin B, Fluconazole, Voriconazole, Anidulafungin, and Caspofungin | Approximately 1 year
  Candida bloodstream isolates were tested for susceptibility to antifungal drugs using the Clinical and Laboratory Standards Institute (CLSI) microbroth dilution method with final readings recorded after 24 hours. The susceptibility cutoffs for antifungal drugs except amphotericin B were from the CLSI M27-S4 Reference Supplement (December 2012). The susceptibility cutoff for amphotericin B was obtained from the published literature.